CLINICAL TRIAL: NCT06234150
Title: Aerobic Dance During Chemotherapy in Breast Cancer Patients With Cognitive Impairment（ADANC）
Brief Title: Aerobic Dance During Chemotherapy in Breast Cancer Patients With Cognitive Impairment
Acronym: ADANC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-SR-732; 2023-SR-732 (Other: Ethics Committee of Nanjing Medical University)
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Neoplasms; Exercise Therapy; Chemotherapy-Related Cognitive Impairment; Cognitive Dysfunction; Dance Therapy
MeSH Terms: conditions — Breast Neoplasms; Chemotherapy-Related Cognitive Impairment; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic dance (Experimental): 50 minutes of moderate-intensity aerobic dance three times a week
  Interventions: Other: Aerobic dance
- Fast-walking (Experimental): 50 minutes of moderate-intensity fast walking three times a week
  Interventions: Other: Fast-walking
- Usual care (No Intervention): Maintain the usual lifestyle and receive medical treatment as normal as the rest of the group.After the baseline evaluation, participants in the control group are asked to maintain their regular lifestyle, including their level of physical activity, and to continue receiving medical treatment and care by standard procedures for 12 weeks. The control group did not receive any encouragement from the researcher to increase the time they spent exercising because, at the time of patient data collection, they were not routinely informed about the benefits of exercise during chemotherapy. Control patients were allowed to engage in the same experimental exercise condition after the 24-week study cycles; if they declined, the study would be stopped.

INTERVENTIONS:
Other: Aerobic dance — Patients assigned to the aerobic dance group will participate in a one-on-one training session before their first chemotherapy session, including aerobic dance instruction, teleconference participation, use of a heart rate bracelet, and use of the Perceived Exertion Rating (PRE) until they master all components. The researchers will also provide participants with instructional videos to view anytime. We will require an exercise log to record the number of workouts, the intensity of the workout using the PRE and heart rate, and the presence of adverse effects. An experienced physical therapist will remotely supervise patients via teleconferencing at home. They will exercise for 50 min three times per week for 12 weeks. The physiotherapist monitors the patient's heart rate throughout the exercise program and provides feedback on any problems encountered during exercise.
  Arms: Aerobic dance
Other: Fast-walking — Patients assigned to the fast-walking group will participate in a one-on-one training session before their first chemotherapy session, including fast-walking instruction, teleconference participation, use of a heart rate bracelet, and use of the Perceived Exertion Rating (PRE) until they master all components. The researchers will also provide participants with instructional videos to view anytime. We will require an exercise log to record the number of workouts, the intensity of the workout using the PRE and heart rate, and the presence of adverse effects. An experienced physical therapist will remotely supervise patients via teleconferencing at home. They will exercise for 50 min three times per week for 12 weeks. The physiotherapist monitors the patient's heart rate throughout the exercise program and provides feedback on any problems encountered during exercise.
  Arms: Fast-walking

SUMMARY:
The goal of this clinical trial is to learn about breast cancer patients. The main questions it aims to answer are:

* Does Aerobic Dance During Chemotherapy Improve Cognitive Function in Breast Cancer Patients？
* Does the efficacy of aerobic dance differ from fast walking of equal intensity？ Recruited patients will be randomly assigned to three groups: (1) aerobic dance group, (2) fast walking group, and (3) usual care group.

The aerobic dance and fast-walking groups participated in supervised exercise lasting 50 minutes thrice a week for 12 weeks.

The goal of this study's findings is to develop practical strategies for managing breast cancer-related cognitive impairment.

DETAILED DESCRIPTION:
BACKGROUND: Cancer-related cognitive impairment (CRCI) is often reported in breast cancer patients and is characterized by a decline in cognitive functions including memory, processing speed, attention, and executive function. Despite the fact that chemotherapy is a significant cause of CRCI, recent studies have shown that 20-30% of patients may already have cognitive decline prior to chemotherapy and that chemotherapy may exacerbate cognitive impairment in these patients. These findings highlight the importance of providing these patients with appropriate interventions while undergoing chemotherapy. A comprehensive form of aerobic exercise known as aerobic dancing has been demonstrated to be effective in alleviating mild cognitive impairment; however, its potential to alleviate cancer-related cognitive impairment is still unknown.

OBJECTIVE: To examine the effects of both aerobic exercises on cognitive function during chemotherapy and compare whether aerobic dance differs from fast walking at the same intensity METHODS: In this three-arm randomized controlled trial, 90 breast cancer patients scheduled for chemotherapy will be randomly assigned to one of three groups: aerobic dance, fast walking, or usual care. The aerobic dance group will participate in three weekly sessions of supervised moderate-intensity exercise, lasting fifty minutes each, for twelve weeks. In contrast, the fast walking group receives the same level of fast-walking intervention, but the usual care group receives no exercise interventions.

RESULTS: The study used the cognitive scales recommended by the International Cognition and Cancer Task Force (ICCTF) with slight modifications for Chinese. The study also included self-reported cognitive function, and assessments on anxiety and depression, quality of life, and sleep. Lymphedema and anthropometry were also included as exploratory indicators.

CONCLUSION: This first-of-its-kind study integrates a novel exercise intervention (Aerobic Dance) with extensive cognitive assessments. If the results are positive, they will serve as a helpful guide for physicians and psychologists to provide women with breast cancer with a comprehensive treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Newly diagnosed, histologically confirmed, resected stage I-IIIa BC
* Scheduled for chemotherapy with Epirubicin+ Cyclophosphamide (EC) regimen
* Presence of objective cognitive decline

Exclusion Criteria:

* Regular exercise habits (exercise at moderate intensity for 30 minutes a day, 3 days a week, for at least 3 months.),
* Motor dysfunction
* Alzheimer's disease
* Vascular dementia

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Shape Trail Test (STT) | From enrollment to the end of treatment at 12 weeks
  Chinese version of the Shape Test (STT-A, STT-B). This test is widely used in China to assess a person's executive function. The Tracking Test (TMT) was created by Partington in 1938. It is divided into two parts, A and B. In part A, the subject must connect 25 numbers on a piece of paper in a specific order; in part B, the subject must connect 25 numbers and letters in alternating order. Since some Chinese may not be familiar with the English alphabet, we used the Chinese version of round and square numbers. The numbers should be connected in sequence, alternating between different shapes. This helps to test the subject's ability to transfer stereotypes, hand-eye coordination, spatial perception and memory. The faster the response, the higher the sensitivity.

SECONDARY OUTCOMES:
the Auditory Word Learning Test - Huashan (AVLT-H) | From enrollment to the end of treatment at 12 weeks
  A scale to test memory function in which the tester reads out 12 words after informing the subject that they need to recall them, and the subject recalls, learns, and recalls the words three times in a row immediately after hearing them, short delayed recall, long-delayed recall, categorical cue recall, and recognition, and the number of words recalled is recorded. Higher scores represent better memory.
Montreal cognitive assessment-basic (MOCA-B) | From enrollment to the end of treatment at 12 weeks
  The Montreal Cognitive Assessment-Basic (MoCA-B) assesses the patient's overall cognitive function. The scale is simple and easy to use and covers several cognitive domains, including attention, executive function, memory, language, visuospatial ability, etc. The higher the score, the better the cognitive function.
Verbal fluency test (VFT) | From enrollment to the end of treatment at 12 weeks
  The number of animal names uttered by the participant within 1 minute is recorded. The more the animal' name is spoken, the better the verbal fluency.
The functional Assessment of Cancer Therapy-Cognitive Function(FACT-Cog) | From enrollment to the end of treatment at 12 weeks
  The Assessment of Cognitive Functioning in Cancer Therapy (FACT-Cog) is a comprehensive scale that assesses self-reported cognitive functioning and consists of the following four sections, Perceived Cognitive Impairment (Cog-PCI), Perceived Cognitive Ability (Cog-PCA), Quality of Life Impacted by Cognitive Impairment (Cog-QoL), and Cognitive Impairment as Perceived by Others (Cog-Oth) for a total of 37 items, with a score of 4 points each. Each item is scored out of 4. The higher the score, the better the self-reported cognitive functioning.
the Functional Assessment of Cancer Therapy-Breast (FACT-B) | From enrollment to the end of treatment at 12 weeks
  Health-related quality of life is assessed using the Functional Assessment of Cancer Therapy-Breast (FACT-B), a 37-item questionnaire designed specifically for breast cancer patients that measures the following five domains: physical, social, emotional, and functional well-being, as well as breast cancer subscales. 3. Sleep quality: assessed using the Pittsburgh Sleep Quality Index, a 19-item questionnaire that assesses seven subjects' sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, sleep medication use, and daytime dysfunction, provides an overall score.
he Hospital Anxiety and Depression Scale（HADS） | From enrollment to the end of treatment at 12 weeks
  a self-report scale usually consisting of 14 entries, of which seven rate depression and seven rate anxiety. It is widely used in studies of psychosomatic disorders and has good reliability and validity. Higher scores indicate severe anxiety-depression symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Cheng Y, Xu L, Xia N, Wang J, Yang W, Jin C, Wang R, Qin J, Zhu Y. Aerobic dance during chemotherapy in patients with breast cancer with cognitive impairment (ADANC): protocol for an assessor-blinded randomised clinical trial. BMJ Open. 2025 Oct 17;15(10):e092003. doi: 10.1136/bmjopen-2024-092003. PMID 41106863